CLINICAL TRIAL: NCT04064255
Title: A Pilot Study Evaluating Practical Body Image (PBI): A Body Image Therapy With Mirror Exposure for Adolescent Inpatients With Anorexia Nervosa
Brief Title: Evaluation of Practical Body Image Therapy for Anorexia Nervosa V1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Newbridge House (Other)
Responsible Party: Principal Investigator, John Morgan, Consultant Psychiatrist, Leeds and York Partnership NHS Foundation Trust
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: NBPBI1992
Record Dates: First submitted 2016-06-23; First posted 2019-08-21 (Actual); Last update posted 2019-08-21 (Actual); Status verified 2019-08

CONDITIONS: Body Image; Exposure
Keywords: Body Image; Anorexia Nervosa; Adolescents; Mirror exposure
MeSH Terms: conditions — Anorexia Nervosa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Case: Practical Body Image + Treatment as Usual (Active Comparator): The Case arm involves Practical Body Image + treatment as usual.
  Practical Body Image is based on a cognitive behavioural model of body image addressing thoughts, feelings, behaviours and misperceptions. PBI is designed to be administered over 10 weeks (6 weekly sessions over 6 weeks, followed by 8 twice weekly sessions over 4 weeks).
  Treatment as usual refers to the standard inpatient treatment programme at Newbridge House which includes: individual therapy, occupational therapy, drama therapy, family therapy, dietetic support, nursing support, yoga and medication prescribed by a consultant psychiatrist.
  Interventions: Other: Practical Body Image (session 1 - 7); Other: Practical Body Image (session 8 - 14)
- Control: Treatment as Usual Only (No Intervention): Control arm involves treatment as usual only.
  Treatment as usual refers to the standard inpatient treatment programme at Newbridge House which includes: individual therapy, occupational therapy, drama therapy, family therapy, dietetic support, nursing support, yoga and medication prescribed by a consultant psychiatrist.

INTERVENTIONS:
Other: Practical Body Image (session 1 - 7) — Practical body image therapy
  Arms: Case: Practical Body Image + Treatment as Usual
Other: Practical Body Image (session 8 - 14) — Twice weekly mirror exposure plus ending session
  Arms: Case: Practical Body Image + Treatment as Usual

SUMMARY:
Background:

Dysfunctional body image is a strong predictor of maintenance and relapse in anorexia nervosa, making treatment of such clinically and financially important. Studies have shown that cognitive behavioural based group therapies and mirror exposure interventions are effective in improving body image in adults with eating disorders; however research into individual body image treatments for adolescents with anorexia nervosa is limited.

Practical Body Image (PBI) is a novel, manualised, individual treatment designed for adolescents with anorexia nervosa for which the evidence base is not yet established. This research will therefore contribute to the evidence base for the treatment of body image in adolescents with anorexia nervosa and inform the effectiveness of a new treatment. The research will be funded by Newbridge House, an inpatient unit for children and adolescents with eating disorders.

Research Questions:

Does Practical Body Image improve body image and psychological wellbeing in adolescent inpatients with anorexia nervosa?

Does a mirror exposure intervention improve body image and psychological wellbeing in adolescent inpatients with anorexia nervosa after completion of the rest of the programme?

Design:

Patients aged 11-18, fulfilling DSM-V criteria for anorexia nervosa and receiving treatment at Newbridge House will be recruited for participation in the research study. Participants will be randomly allocated to either a case or control group. Allocation will be based on a non-blind randomised controlled trial. Cases will receive PBI in addition to treatment as usual and will be compared with controls who just receive treatment as usual. Both groups will complete a set of questionnaires at baseline, 7 weeks and 10 weeks.

DETAILED DESCRIPTION:
PRINCIPAL NULL HYPOTHESIS PBI will have no impact on body image or psychological wellbeing in adolescent inpatients with anorexia nervosa compared to just TAU.

SECONDARY NULL HYPOTHESIS Mirror exposure will have no effect on body image or psychological wellbeing in adolescent inpatients with anorexia nervosa after completion of the rest of PBI.

PRINCIPAL ALTERNATIVE HYPOTHESIS PBI will improve body image and psychological wellbeing in adolescent inpatients with anorexia nervosa compared to just TAU.

SECONDARY ALTERNATIVE HYPOTHESIS Mirror exposure will improve body image and psychological wellbeing in adolescent inpatients with anorexia nervosa after completion of the rest of PBI.

The alternative hypotheses were chosen based previous research which shows that cognitive behavioural techniques and mirror exposure are effective in improving body image disturbance and psychological wellbeing in adults with anorexia nervosa. This study aims to generate hypotheses about which specific elements of body image (i.e. body avoidance, body acceptance, body anxiety or weight and shape concern) and psychological wellbeing (i.e. self esteem, anxiety and depression) change after completion of PBI.

DESIGN

The principal hypothesis will be tested using a between subjects design (PBI vs no PBI) with treatment as the independent variable. The case group will receive TAU as well as PBI and the control group will receive just TAU. The outcomes from self-report measures completed at 10 weeks will be compared between the case and control groups to answer the principal research question.

The secondary hypothesis will be tested using a within subjects design (before mirror exposure vs after mirror exposure) with mirror exposure as the independent variable. The case group will complete self-report measures at week 7 before commencing mirror exposure in addition to week 10. This will allow comparison of outcomes before mirror exposure to after mirror exposure to answer the secondary research question.

The dependent variables are body image (including body avoidance, acceptance, anxiety and weight and shape concerns) and psychological wellbeing (including self-esteem, anxiety and depression) as measured by self-report questionnaires.

This experimental design has been chosen as it allows for the comparison of PBI vs no PBI as well as a comparison between outcomes before mirror exposure and outcomes after mirror exposure. The choice of this design was influenced by a desire to provide an evidence base for this novel treatment and to determine whether mirror exposure has any additional benefit for adolescents with anorexia nervosa.

METHOD

Participants will be inpatients, aged 11 - 18, fulfilling DSM-IV criteria for anorexia nervosa and receiving treatment at Newbridge House child and adolescent inpatient eating disorder unit. A convenience sampling method will be used and participants will be randomly allocated to either a 'case' group to complete TAU plus PBI or a 'control' group to complete only TAU using an Excel formula. A control group (TAU) was included in order to compare outcomes of those who complete PBI with outcomes of those who do not. This is because the principal aim of the study is to evaluate the effectiveness of this novel treatment and there is insufficient evidence to support the introduction of PBI without conducting a study of this kind. This is especially necessary given that the research site is an inpatient unit and all participants will be receiving other therapies alongside the treatment being tested.

Forty participants will be recruited in total (twenty in each group). As this is a pilot study no power calculation could be conducted and this sample size was agreed as sufficient to generate data to inform a power calculation for future research. Participants will be identifiable by a unique code created using the letters 'TAU+PBI' or 'TAU' followed by a number relating to the order in which they were recruited (1-20). Participants will be approached to take part in the research when they reach 90% of their healthy weight. All patients on the unit who fulfill the framework of inclusion and exclusion criteria will be asked for their informed written consent to participate after reading a research information sheet. For patients under age 16, parents will also be given a research information sheet and consent form and asked to provide written informed consent.

TIMETABLE

All stages will take place on site at Newbridge House.

STAGE 0 (Recruitment)

Patients will be recruited as described above and an Assistant Psychologist will meet with them to read through the research information sheet and request informed written consent. For patients under 16, written parental consent will also be sought and parents will be given an information sheet and consent form prior to commencement of the study. Patients and parents will be given 7 days to consider their decision to consent to participate in the research. Patients for whom we receive consent will then be randomly allocated to either the case or control group using an Excel formula. Patients who do not consent, or for whom parental consent is not received, will not be included in the study and will receive TAU which will be identical to that delivered to controls. Patients declining to participate will be asked for permission to use demographic and routine clinical data to test if there are any significant differences between participants versus non-participants, and to examine whether the sample is representative.

Stage 1 (Week 1)

All participants will be asked to complete a set of self-report measures in week 1 (baseline). For participants in the case group, PBI will then commence and take place over 7 weeks alongside TAU. For participants in the control group TAU will continue.

STAGE 2 (Week 7)

Stage 2 will take place 7 weeks after completion of baseline measures in between session 7 and 8 of PBI. At this stage the same measures will be completed by participants in the case group only.

For participants in the case group, the mirror exposure part of PBI will commence and take place twice a week, over 3 weeks alongside TAU. For participants in the control group TAU will continue.

STAGE 3 (Week 10)

Stage 3 will take place 10 weeks after completion of baseline measures. At this stage those in the case group will have completed the PBI intervention. The same measures will be completed for the last time by participants in both the case and control groups.

Participant feedback about their experiences of the programme will also be sought.

STAGE 4 (Data analysis)

Researchers will input raw data from completed outcome measures onto an SPSS spreadsheet. Data will then be analysed and interpreted.

STAGE 5 (Report write up)

The final report will be written for publication.

INTERVENTION The intervention will comprise of 14 sessions of individual body image therapy using a cognitive behavioural approach over a 10 week period. The therapy has been protocolised into a treatment manual known as PBI, and will be administered by Assistant Psychologists employed at Newbridge House receiving weekly supervision from a Clinical Psychologist.

PBI is based on a cognitive behavioural model of body image addressing thoughts, feelings, behaviours and misperceptions. PBI is designed to be administered over 6 weekly sessions followed by 8 twice weekly sessions over 4 weeks. Therapists delivering the programme will have time to read through the manual and attend weekly peer supervision to support adherence to the protocol. Therapists will require some background knowledge of the nature of body image in eating disorders and some knowledge of basic CBT principles. They will also receive weekly clinical supervision by a trained CBT therapist. The sessions are structured and laid out in the following overview:

Week 1, Session 1: My Body Image

Week 2, Session 2: Body Perception

Week 3, Session 3: Testing Beliefs

Week 4, Session 4: Body Avoidance Outing 1

Week 5, Session 5: Body Avoidance Outing 2

Week 6, Session 6: Review and Reflection

Week 7, Session 7: Introduction to Mirror Use Session 8: Mirror Exposure 1

Week 8, Session 9: Mirror Exposure 2 Session 10: Mirror Exposure 3

Week 9, Session 11: Mirror Exposure 4 Session 12: Mirror Exposure 5

Week 10,Session 13: Mirror Exposure 6 Session 14: Ending Session

Week 10, Session 13: Mirror Exposure, Session 14: Ending session

ELIGIBILITY:
Inclusion Criteria:

1. Inpatients at Newbridge House
2. Aged 11-18
3. At or above 90% of minimum healthy weight
4. Primary diagnosis of Anorexia Nervosa

Exclusion Criteria:

1. Previously received treatment at Newbridge House (readmission)
2. Patients with a primary diagnosis other than Anorexia Nervosa
3. Aged under 11 years
4. Any patients with severe learning difficulty
5. Active psychosis

Ages: 11 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2018-07 (Actual); Study Completion 2018-07-01 (Actual)

PRIMARY OUTCOMES:
Body Image Acceptance and Action Questionnaire | Assessed at baseline, 7 weeks and 10 weeks.
  A validated self-report measure assessing change in cognitive flexibility and acceptance relatively to body image. The measure consists of 12 questions.

SECONDARY OUTCOMES:
Youth Eating Disorder Examination Questionnaire | Assessed at baseline, 7 weeks and 10 weeks.
  This is the youth version of the EDE-Q which is a validated self-report measure assessing change in eating disorder psychopathology using four sub-scales measuring weight concern, shape concern, dietary restraint and eating concern. The measure consists of 39 questions.
Body Image Avoidance Questionnaire | Assessed at baseline, 7 weeks and 10 weeks.
  A validated self-report measure assessing change in body image avoidance divided into three sub-scales including social avoidance, clothing avoidance and personal grooming. The measure consists of 12 questions.
Physical Appearance State and Trait Anxiety Scale: Trait Version | Assessed at baseline, 7 weeks and 10 weeks.
  A validated self-report measure assessing change in trait anxiety relating to physical appearance. The measure consists of 16 questions.
Healthy weight body acceptance scale | Assessed at baseline, 7 weeks and 10 weeks.
  A non validated self-report measure assessing change in what having a healthy weight body means to a person, acceptance of having a healthy weight body and the motivation and confidence to accept having a healthy weight body. The measure consists of 4 questions.

CONTACTS AND LOCATIONS:
Overall Officials: John F Morgan, Medicine, Principal Investigator — Yorkshire Centre for Eating Disorders, Leeds and York NHS Foundation Trust

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stice E. Risk and maintenance factors for eating pathology: a meta-analytic review. Psychol Bull. 2002 Sep;128(5):825-48. doi: 10.1037/0033-2909.128.5.825. PMID 12206196
- [Background] Fairburn CG, Peveler RC, Jones R, Hope RA, Doll HA. Predictors of 12-month outcome in bulimia nervosa and the influence of attitudes to shape and weight. J Consult Clin Psychol. 1993 Aug;61(4):696-8. doi: 10.1037//0022-006x.61.4.696. PMID 8370866
- [Background] Keel PK, Dorer DJ, Franko DL, Jackson SC, Herzog DB. Postremission predictors of relapse in women with eating disorders. Am J Psychiatry. 2005 Dec;162(12):2263-8. doi: 10.1176/appi.ajp.162.12.2263. PMID 16330589
- [Background] Morgan JF, Lazarova S, Schelhase M, Saeidi S. Ten session body image therapy: efficacy of a manualised body image therapy. Eur Eat Disord Rev. 2014 Jan;22(1):66-71. doi: 10.1002/erv.2249. Epub 2013 Sep 5. PMID 24006359
- [Background] Key A, George CL, Beattie D, Stammers K, Lacey H, Waller G. Body image treatment within an inpatient program for anorexia nervosa: the role of mirror exposure in the desensitization process. Int J Eat Disord. 2002 Mar;31(2):185-90. doi: 10.1002/eat.10027. PMID 11920979
- [Background] Legenbauer T, Schutt-Stromel S, Hiller W, Vocks S. Predictors of improved eating behaviour following body image therapy: a pilot study. Eur Eat Disord Rev. 2011 Mar-Apr;19(2):129-37. doi: 10.1002/erv.1017. PMID 25363718
- [Background] Nye S, Cash TF. Outcomes of manualized cognitive-behavioral body image therapy with eating disordered women treated in a private clinical practice. Eat Disord. 2006 Jan-Feb;14(1):31-40. doi: 10.1080/10640260500403840. PMID 16757447
- [Background] Delinsky SS, Wilson GT. Mirror exposure for the treatment of body image disturbance. Int J Eat Disord. 2006 Mar;39(2):108-16. doi: 10.1002/eat.20207. PMID 16231342